CLINICAL TRIAL: NCT01412814
Title: Biomechanics of Gait Pattern Adaptation in Patients After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC 11 MS 0569-10-TLV CTIL; 0569-10-TLV (Registry Identifier: Institutional Review Board Sourasky Medical Center)
Record Dates: First submitted 2011-07-20; First posted 2011-08-09 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Knee Arthroplasty; Knee Arthritis Osteoarthritis; Osteoarthritis; Osteoarthritis, Knee; Musculoskeletal Diseases
Keywords: Total knee arthroplasty; Total knee replacement; End-stage knee osteoarthritis; Gait patterns; Neuromuscular education
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Experimental (Experimental): These patients will carry out the specified intervention of the study with the AposTherapy Biomechanical System in addition to the typical physical therapy regiment prescribed to them by their physician.
  Interventions: Device: AposTherapy Biomechanical System
- Control (Active Comparator): The patients within this group will also carry out the typical physical therapy program for total knee replacement as prescribed by their physician. The patients will carry out a similar therapy program to the experimental group, but without the study intervention device (placebo walking shoe).
  Interventions: Other: Physical Therapy Program

INTERVENTIONS:
Device: AposTherapy Biomechanical System — The device is comprised of four adjustable modular elements attached to foot-worn platforms that are capable of manipulating the foot's center-of-pressure and applying perturbation training throughout the gait cycle. The device allows for neuromuscular training during dynamic loading.
  Arms: Experimental
Other: Physical Therapy Program — Their therapy program will be similar to the experimental group, but without the treatment device (placebo walking shoe).
  Arms: Control

SUMMARY:
This study aimed to discover the biomechanics of gait pattern adaptation in patients after a total knee replacement.

The first hypothesis of the project was that center-of-pressure manipulation at the foot during dynamic loading is capable of changing the forces, torques and muscle activation patterns of the lower limb.

The second hypothesis of the project was that patient-specific center-of-pressure manipulation at the foot combined with repetitive perturbation training over time will improve neuromuscular function, barefoot gait patterns, muscle activation patterns, pain, quality of life and energy consumption in patients after a total knee replacement.

DETAILED DESCRIPTION:
This study is a randomized prospective controlled study of patients after total knee arthroplasty. Patients will be recruited to the study and divided randomly into an experimental and control group. Both groups will match in terms of gender, age, pathology and clinical assessment. In addition to the intervention of the present study, all patients, whether in the experimental or control group, will carry out the usual physical therapy exercises for total knee arthroplasty as directed by their physician. The patients will be recruited and evaluated prior to surgery and for a follow-up period after surgery.

After surgery, patients in the experimental group will be fitted with a customized biomechanical device worn on the feet (Apos System, Apos - Sports and Medical Technologies Ltd. Hertzlia, Israel). The device is calibrated personally to each patient. By calibrating the device, the center-of-pressure of the foot can be manipulated during all phases of the gait cycle. The device is capable of inducing controlled perturbation during gait. The immediate effects of the device will be evaluated using center-of-pressure measurements, three-dimensional gait analyses and surface electromyography. The patients are instructed to walk with the device according to a therapy protocol (AposTherapy). Patients will be evaluated for changes in gait via three-dimensional gait analyses, muscle activation pattern changes via surface electromyography, pain, quality of life and energy consumption.

The patients in the control group will carry out the same walking exercises as the experimental group, but without the biomechanical intervention device (placebo walking shoe). The patients will be evaluated with the same tools over time as with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for first total knee arthroplasty due to end-stage knee osteoarthritis
* Ambulatory and active patients that can participate in gait analysis

Exclusion Criteria:

* Prior joint surgery of either lower extremity, with the exception of arthroscopy
* Unsteady gait
* Back pain
* Neurological, pulmonary or cardiovascular pathologies or risks that may affect long-term performance
* Inability to understand or comply with the treatment protocol

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Gait Patterns at 6-8 weeks, 5-6 months and 11-12 months | An average of 2 weeks prior to surgery and an average of 6-8 weeks, 5-6 months and 11-12 months after surgery
  Three-dimensional gait analysis of spatiotemporal, kinetic and kinematic parameters.
  Surface electromyographic analysis of muscle activation patterns. Center of pressure measurements and function tests.

SECONDARY OUTCOMES:
Change from Baseline in Pain, Function and Quality of Life Assessments at 6-8 weeks, 5-6 months and 11-12 months | An average of 2 weeks prior to surgery and an average of 6-8 weeks, 5-6 months and 11-12 months after surgery
  Includes self-evaluation questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Biorobotics and Biomechanics Lab, Technion Israel Institute of Technology, Haifa, Israel, Israel